CLINICAL TRIAL: NCT06134843
Title: A Single-Blind, Randomized, Controlled, Single Center Clinical Study to Assess the Safety and Efficacy of DERMASEAL Advanced Wound Care Dressing for the Treatment of Split-Thickness Skin Graft Donor Site Wounds
Brief Title: Study to Assess the Safety and Efficacy of DERMASEAL for the Treatment of Split-Thickness Skin Graft Donor Site Wounds
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hobart W. Harris (Industry)
Collaborators: Vitruvian Medical Devices, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Hobart W. Harris, President, Vitruvian Medical Devices, Inc.
Organization: Vitruvian Medical Devices, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VMD2022-002
Record Dates: First submitted 2023-11-04; First posted 2023-11-18 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Skin Graft Complications
Keywords: pain; scarring; wound healing
MeSH Terms: conditions — Pain; Cicatrix

STUDY DESIGN:
Intervention Model Description: single center, single-blind, randomized, controlled interventional study
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessors will evaluate pain and scarring using the Visual Analog Scale (VAS) Vancouver Scar Scale (VSS) without knowledge of the participants' treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DERMASEAL (Experimental): DERMASEAL will be placed to completely cover the donor site wound. The entire site will then be covered with a transparent film dressing (TegadermTM, 3M) with at least 3 cm margin of normal skin under the film dressing before securing it with kerlix gauze and an ace wrap bandage placed circumferentially around the extremity.
  The dressing will be left on the donor site wound until the wound is completely closed or changed at the discretion of the treating team.
  Interventions: Combination Product: DERMASEAL
- Standard of Care (No Intervention): The donor site wound is covered with a transparent film dressing (TegadermTM, 3M) with at least 3 cm margin of normal skin under the film dressing. The dressing is then secured with kerlix gauze and ace wrap bandage placed circumferentially around the extremity.
  The dressing will be left on the donor site wound until the wound is completely closed or changed at the discretion of the treating team.

INTERVENTIONS:
Combination Product: DERMASEAL — plasma film containing metallic silver microparticles and fibrin
  Arms: DERMASEAL

SUMMARY:
The goal of this study to determine whether the combination biologic/drug DERMASEAL will safely decrease donor wound pain after split-thickness skin graft surgery. Participants will have their skin graft donor sites immediately treated with DERMASEAL versus standard of care wound dressings followed by periodic monitoring of their recovery.

DETAILED DESCRIPTION:
This is a single center, single-blind, randomized, controlled phase 1/2 study of patients undergoing treatment of a cutaneous wound involving a split-thickness skin graft. A subject's study duration will be for up to a total of 16 weeks from randomization to end of study. This includes 1 week of treatment, followed by 3 weeks of Standard of Care plus a final follow-up visit 12 weeks after complete wound closure or the end of Standard of Care.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 21 years of age.
2. The subject is able and willing to adhere to study procedures and informed consent is obtained.
3. Patient scheduled to undergo a split-thickness skin graft > 25 cm2 and ≤ 300 cm2 with a wound depth of between 0.010 - 0.015 inch (0.2 - 0.4 mm).
4. Target donor site wound involving the torso or upper or lower extremities.
5. Patient has a palpable pulse at the wrist or ankle indicating adequate arterial perfusion of the extremity from which the skin graft is harvested.
6. Serum creatinine <2.0 mg/dl within the last 6 months.
7. Negative urine pregnancy test at screening for women of childbearing potential. i) Women participants are considered of non-childbearing potential if they are pre-menopausal with a documented hysterectomy or bilateral oophorectomy; or post-menopausal defined as the cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; or have a serum FSH level confirming the post-menopausal state.

Exclusion Criteria:

1. Hypersensitivity to silver or fresh frozen plasma.
2. Active infection or history of radiation to the donor site.
3. Insensate at the donor site.
4. Elevated INR>3.0.
5. The subject was previously entered into this study or had participated in any study drug or medical device study within 30 days of screening.
6. Currently on a treatment regimen or medications which in the opinion of the investigator are known to interfere with wound healing (for example: cancer chemotherapy or equivalent immunosuppressants, systemic steroids > 10 days of treatment, cytostatic drugs, COX-2 inhibitors, or radiation therapy).
7. Excessive lymphedema that in the opinion of the investigator will interfere with wound healing.
8. A cognitive, physical, or psychological condition interfering with subject's ability to comply with the treatment regimen.
9. Subject is on dialysis.
10. Patients who are pregnant, breast feeding, or unwilling to practice contraceptive methods during participation in the study, if applicable. Effective methods of contraception include:

    i. oral, injectable, or implanted hormonal contraceptives ii. intrauterine device or system, iii. barrier method with spermicide, or iv. bilateral tubal occlusion.
11. Patients with uncontrolled anemia (Hgb<10 g/dL in women; <12 g/dL in men) at Screening.
12. Severe malnutrition (serum albumin ≤2.0 with a normal CRP).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
adverse events | 16 weeks
  The safety of topically applying a plasma film containing metallic silver microparticles plus fibrin in patients with skin graft donor sites for 16 weeks following split-thickness skin grafting.
wound pain | 16 weeks
  The study will evaluate if using DERMASEAL is associated with a clinically meaningful difference in pain score (≥2 points on the Visual Analog Scale; minimal score =0 and maximal score = 10. A higher score means more pain) between the treatment and active control arms at any time during the 16-week study.

SECONDARY OUTCOMES:
Percent wound healing | 4 weeks
  Percent of donor site wounds healed during the post-treatment weeks 1 through 4
Time to complete wound closure | 4 weeks
  Time to complete donor site wound closure during the post-treatment weeks 1 through 4
Recurrent donor site wound after complete wound closure | 16 weeks
  Recurrence of donor site after complete wound closure, requiring treatment, at any time during the 16-week study.
Scarring | 16 weeks
  Scarring as measured by the Vancouver Scar Scale at 16 weeks after surgery. The minimum value = 0 and maximal value = 13; higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David M Young, MD, Principal Investigator — UCSF School of Medicine

IPD SHARING:
Plan to Share IPD: No